CLINICAL TRIAL: NCT05105698
Title: Food-effect Bioavailability of Gemigliptin and Dapagliflozin 50/10 mg Fixed Dose Combination Film-coated Tablet Under Fed and Fasting Conditions in Healthy Volunteers
Brief Title: Food-effect Bioavailability of Gemigliptin and Dapagliflozin 50/10 mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GLCL003
Record Dates: First submitted 2021-10-13; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LC15-0444; dapagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fasting conditions (Experimental): A: A fixed dose combination of gemigliptin and dapagliflozin 50/10 mg film-coated tablet orally administered once without food (fasting conditions)
  Interventions: Drug: gemigliptin and dapagliflozin 50/10 mg film-coated tablet (Fasting)
- fed conditions (Experimental): B: A fixed dose combination of gemigliptin and dapagliflozin 50/10 mg film-coated tablet orally administered once with food (fed conditions)
  Interventions: Drug: gemigliptin and dapagliflozin 50/10 mg film-coated tablet (fed)

INTERVENTIONS:
Drug: gemigliptin and dapagliflozin 50/10 mg film-coated tablet (Fasting) — Subjects will check-in a night before investigational product administration, supervised for at least 8 hours overnight fasting prior to dosing and in-house stay until 24 hours post-dose.(fasting)
  Other Names: DPP-4 inhibitor and SGLT-2 inhibitor combination
  Arms: fasting conditions
Drug: gemigliptin and dapagliflozin 50/10 mg film-coated tablet (fed) — Subjects will check-in a night before investigational product administration, supervised for at least 8 hours overnight fasting prior to dosing and in-house stay until 24 hours post-dose.(fed)
  Other Names: DPP-4 inhibitor and SGLT-2 inhibitor combination
  Arms: fed conditions

SUMMARY:
A Randomized, Open-label, Single-dose, Two-way Crossover Study to Investigate Food-effect Bioavailability of Gemigliptin and Dapagliflozin 50/10 mg Fixed Dose Combination Film-coated Tablet under Fed and Fasting Conditions in Healthy Volunteers

DETAILED DESCRIPTION:
[Objectives]

* Primary: To investigate the food-effect bioavailability of absorption of gemigliptin and dapagliflozin 50/10 mg fixed dose combination film-coated tablet in healthy subjects under fed and fasting conditions
* Secondary: To evaluate safety of investigational product under fed and fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Male and female, healthy volunteers aged 18-55 years, body mass index between 18.0 to 30.0 kg/m2. All of them should be able to complete the clinical study including the follow-up and capable of providing written informed consent.

Exclusion Criteria:

* History serious hypersensitivity reactions
* History or evidence of clinically significant renal, hepatic, gastrointestinal
* Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19
* History about administration of first dose or second dose of COVID-19 vaccine within 30 days prior to check-in in each Period
* History or evidence of family diabetes
* History or evidence of type 1 diabetes mellitus, diabetic ketoacidosis, diabetic pre-coma
* etc.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Blood samples will be collected at time 0.00 and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00,12.00, 24.00, 48.00
  Cmax will be determined from the plasma concentration data of gemigliptin, LC15-0636 and dapagliflozin
Area under the plasma concentrationup up to the last measurable concentration (AUC0-tlast) | Blood samples will be collected at time 0.00 and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00,12.00, 24.00, 48.00
  AUC0-tlast will be determined from the plasma concentration data of gemigliptin, LC15-0636 and dapagliflozin
Area under the plasma concentration-time curve to from time 0 to infinite(AUC0-∞) | Blood samples will be collected at time 0.00 and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00,12.00, 24.00, 48.00
  AUC0-∞ will be determined from the plasma concentration data of gemigliptin, LC15-0636 and dapagliflozin

IPD SHARING:
Plan to Share IPD: No